CLINICAL TRIAL: NCT00560508
Title: A Double-blind, Double-dummy, Randomised, Parallel-group Study to Investigate the Safety, Tolerability, Trough Plasma Concentration, and Efficacy of Pramipexole ER Versus Pramipexole Immediate Release (IR) Administered Orally for 12 Weeks in Patients With Parkinson's Disease (PD) on L-dopa Therapy, Followed by a 52-week Open-label Long-term Treatment Period to Evaluate the Long-term Safety and Efficacy of Pramipexole ER
Brief Title: A 12-week Study of Pramipexole Extended Release (ER) in Patients With Parkinson's Disease (PD), Followed by a 52-week Long-term Treatment Period
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.610
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pramipexole Extended Release (Experimental): patient to receive a tablet containing 0.375 mg Pramipexole ER once a day plus containing 0.125 mg Pramipexole IR placebo twice a day -> a tablet containing 1.5 mg Pramipexole ER three times daily (TID) plus 0.5 mg Pramipexole IR placebo TID
  Interventions: Drug: Pramipexole Extended Release
- Pramipexole Immediate Release (Active Comparator): patient to receive a tablet containing 0.125 mg Pramipexole IR twice a day plus containing 0.375 mg Pramipexole ER placebo once a day -> a tablet containing 0.5 mg Pramipexole IR three times daily (TID) plus 1.5 mg Pramipexole ER placebo TID
  Interventions: Drug: Pramipexole Immediate Release

INTERVENTIONS:
Drug: Pramipexole Immediate Release — titrated as individually needed (0.25 mg - 4.5 mg daily)
  Arms: Pramipexole Immediate Release
Drug: Pramipexole Extended Release — titration as individually needed (0.375 mg -4.5 mg daily)
  Arms: Pramipexole Extended Release

SUMMARY:
The objective of this trial is to investigate the safety, tolerability, trough plasma concentration, and efficacy of pramipexole ER in comparison with those of pramipexole IR administrated orally for 12 weeks in patients with PD on levodopa (L-DOPA) therapy (the double-blind period). The double-blind period will be followed by the open-label 52 week administration of pramipexole ER to evaluate the long term safety and efficacy (the open-label period).

ELIGIBILITY:
Inclusion criteria

1. Male or female patients with diagnosis of PD including juvenile Parkinsonism, in whom the onset began at the age of forty or younger.
2. Patients with a modified Hoehn and Yahr scale of II to IV at "on" time.
3. Patients who have received an individual dosage of L-DOPA (either standard L-DOPA or L-DOPA with dopa-decarboxylase inhibitor) at a stable dose for at least 4 weeks before the baseline visit (Visit 2).
4. Patients who exhibit any therapeutically problematic issues or status based on L-DOPA therapy:

   * wearing-off phenomena
   * no on /delayed on
   * dystonia at off time
   * on-off phenomena
   * freezing phenomena at off time
   * the sub-optimal dose of L-DOPA had been administered due to side effects (such as dyskinesia), or therapeutical strategy

Exclusion criteria

1. Atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases.
2. Dementia, as defined by a Mini-Mental State Examination (MMSE) score <24 at screening visit.
3. Any psychiatric disorder according to DSM-IV criteria that could prevent compliance or completion of the trial and/or put the patient at risk if he/she takes part in the trial.
4. History of psychosis, except history of drug induced hallucinations (provided the investigator considers that participation in the trial would not represent a significant risk for the patient).
5. Clinically significant ECG abnormalities at screening visit, according to investigator's judgement.
6. Clinically significant hypotension or symptomatic orthostatic hypotension (i.e., clinical symptoms of orthostatic hypotension such as dizziness postural etc associated with a decline >=20 mmHg in systolic blood pressure and a decline >=10 mmHg in diastolic blood pressure, at one minute after standing compared with the previous supine systolic and diastolic blood pressure obtained after 5 minutes of quiet rest) either at screening visit or at baseline visit.
7. Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the trial.
8. Pregnancy (to be excluded by serum pregnancy test at screening visit) or breast-feeding.
9. Sexually active female of childbearing potential not using a medically approved method of birth control within one month before to the screening visit and throughout the trial period.
10. Serum levels of AST, ALT, alkaline phosphatases or bilirubin >2 upper limits of normal .
11. Patients with a creatinine clearance <50 mL/min
12. Patients with a complication or signs of malignant tumours or those within 5 years after the treatment.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- Japan (19):
  - 248.610.019 Boehringer Ingelheim Investigational Site, Akashi, Hyogo
  - 248.610.020 Boehringer Ingelheim Investigational Site, Akita, Akita
  - 248.610.006 Boehringer Ingelheim Investigational Site, Aomori, Aomori
  - 248.610.017 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 248.610.018 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 248.610.001 Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - 248.610.014 Boehringer Ingelheim Investigational Site, Fuchu, Tokyo
  - 248.610.011 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 248.610.015 Boehringer Ingelheim Investigational Site, Iwamizawa,Hokkaido
  - 248.610.003 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 248.610.008 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 248.610.021 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 248.610.010 Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - 248.610.005 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 248.610.012 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 248.610.004 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 248.610.009 Boehringer Ingelheim Investigational Site, Shimogyo-ku, Kyoto, Kyoto
  - 248.610.007 Boehringer Ingelheim Investigational Site, Shiroishi, Miyagi
  - 248.610.002 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole Extended Release Group (PPX ER): Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day
- Pramipexole Immediate Release Group (PPX IR): Pramipexole Immediate Release (IR) tablets of 0.125 mg and 0.5 mg dose: 0.25 mg, 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg, 2.5 mg, 3.0 mg, 3.5 mg, or 4.5 mg, twice or three times a day
Period: 12 Week Double-blind Period
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Started | 56 | 56
Completed | 51 | 53
Not Completed | 5 | 3
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: 52-week Open-label Period Pramipexole ER
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Started | 51 (all patients received Pramipexole ER for the 52-week open-label period) | 53 (all patients received Pramipexole ER for the 52-week open-label period)
Completed | 43 | 42
Not Completed | 8 | 11
Not completed — Adverse Event | 6 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other reason - investigator's judgement | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pramipexole Immediate Release Group (PPX IR): Pramipexole IR (tablets of 0.125 mg and 0.5 mg) dose: 0.25 mg, 0.5 mg, 1.0 mg, 1.5 mg, 2.0 mg, 2.5 mg, 3.0 mg, 3.5 mg, or 4.5 mg, twice or three times a day
- Total: Total of all reporting groups
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR) | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (8.0) | 66.1 (7.5) | 67.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 21 | 21 | 42

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Parts II+III Total Score
Description: UPDRS II+III ranging from 0 point(normal) to 160 point (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
UPDRS scores on a scale | -13.6 (1.3) | -13.3 (1.3)

2. Secondary Outcome: Change From Baseline in Percentage Off-time
Description: Percentage off-time during waking hours in the last two days based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease).
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage of off-time
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
Percentage of off-time | -5.8 (2.4) | -7.8 (2.4)

3. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia
Description: Percentage on-time without dyskinesia during waking hours in the last two days based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
Percentage of on-time | 6.4 (2.5) | 7.0 (2.5)

4. Secondary Outcome: Change From Baseline in Percentage On-time With Non-troublesome Dyskinesia
Description: Percentage on-time with non-troublesome dyskinesia during waking hours in the last two days based on patient diary data, percentage ranging from 0(worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
Percentage of on-time | -0.4 (0.4) | 0.1 (0.4)

5. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia or With Non-troublesome Dyskinesia
Description: Percentage on-time without dyskinesia or non-troublesome dyskinesia during waking hours in the last two days based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
Percentage of on-time | 6.0 (2.5) | 7.1 (2.5)

6. Secondary Outcome: Change From Baseline in Percentage On-time With Troublesome Dyskinesia
Description: Percentage on-time with troublesome dyskinesia during waking hours in the last two days based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
Percentage of on-time | -0.1 (0.5) | 0.5 (0.5)

7. Secondary Outcome: Responder Rate For Clinical Global Impression of Improvement (CGI-I)
Description: CGI-I scores ranging from '1' (very much improved) to '7' (very much worse), CGI-I responder have scoring of 1 or 2 (at least much improved)
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
percentage of participants | 48.2 | 50.0

8. Secondary Outcome: Responder Rate For Patient Global Impression of Improvement (PGI-I)
Description: PGI-I scores ranging from '1' (very much better) to '7' (very much worse), PGI-I responder have scoring of 1 or 2 (at least much better)
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
percentage of participants | 33.9 | 33.9

9. Secondary Outcome: Change From Baseline in UPDRS Part I Score
Description: UPDRS Part I ranging from 0 (normal) to 16 (severe). UPDRS Part I measures Mentation, Behavior and Mood
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
UPDRS scores on a scale | 0.1 (0.2) | -0.2 (0.2)

10. Secondary Outcome: Change From Baseline in UPDRS Part II Score
Description: UPDRS Part II ranging from 0 (normal) to 52 (severe). UPDRS Part II is calculated as the average of UPDRS Part II at on and UPDRS Part II at off-period for each of the 13 activities.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
UPDRS scores on a scale | -3.3 (0.4) | -3.4 (0.4)

11. Secondary Outcome: Change From Baseline in UPDRS Part III Score
Description: UPDRS Part III ranging from 0 (normal) to 108 (severe). UPDRS Part III measures motor symptoms
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
UPDRS scores on a scale | -10.2 (1.0) | -9.9 (1.0)

12. Secondary Outcome: Change From Baseline in UPDRS Part IV Score
Description: UPDRS Part IV ranging from 0 (normal) to 23 (severe). UPDRS Part IV measures complications of therapy
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
UPDRS scores on a scale | -0.2 (0.2) | -0.4 (0.2)

13. Secondary Outcome: UPDRS Parts II+III Total Score Responder Rate (at Least 20% Improvement)
Description: Responders are defined as at least 20% decrease in the UPDRS Parts II+III Total Score ranges 0-160 scores from best to worse
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
percentage of participants | 78.6 | 82.1

14. Secondary Outcome: Change From Baseline in L-dopa Daily Dose
Description: The L-dopa daily dose was recorded in the electronic case report form (eCRF) at each trial visit.
Time Frame: baseline and after 12 weeks treatment
Population: Full Analysis Set (FAS) with last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mg per day
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
mg per day | -5.3 (3.0) | -1.8 (3.0)

15. Primary Outcome: Percentage of Participants Who Experienced Adverse Events
Description: An adverse event is defined as any untoward medical occurrence
Time Frame: 12 weeks
Population: Treated set for safety, which was the analysis set including all the patients who had valid measurements after drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 56 | 56
percentage of participants | 83.93 | 83.93

16. Secondary Outcome: Trough Plasma Concentration at Steady State
Description: Geometric mean (gMean) was calculated for trough plasma concentrations of pramipexole at steady state after administration of pramipexole IR 4.5mg and pramipexole ER 4.5mg.
Time Frame: at Visit 8 after pramipexole ER 4.5mg and IR 4.5mg treatment
Population: Full Analysis Set (FAS)
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Number analyzed (Participants) | 24 | 30
ng/ml | 5.46 (2.01) | 5.09 (2.53)

17. Secondary Outcome: Dose Proportionality of Trough Plasma Concentration at Steady State After Pramipexole ER Treatment
Description: Dose proportionality of trough plasma concentrations at steady state is explored by using the power model that described the functional relationship between the dose and plasma concentration
Time Frame: from Visit 1 to Visit 8 after pramipexole ER
Population: Full Analysis Set (FAS).
Measure: Mean (Standard Error); unit: ng/mL
Units Other Than Participants: Cpre,ss (ng/ml) for Pramipexole (Plasma)
Arm/Group | Pramipexole Extended Release Group (PPX ER)
Number analyzed (Participants) | 56
Number analyzed (Cpre,ss (ng/ml) for Pramipexole (Plasma)) | 195
ng/mL | 1.0375 (0.0177)

18. Secondary Outcome: Change From End of Double-Blind Period in UPDRS (Unified Parkinson's Disease Rating Scale) Parts II+III Total Score (Open-label: Dose Adjustment Phase)
Description: UPDRS II+III ranging from 0 point(normal) to 160 point (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms. Least square means and standard errors presented are from ANCOVA with factors treatment and covariate baseline.
Time Frame: Week 12 to Week 16
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Groups:
- From PPX ER to PPX ER: Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day
- From PPX IR to PPX ER: From Pramipexole IR (tablets of 0.125 mg and 0.5 mg) dose: 0.25 mg, 1.0 mg, 1.5 mg, 2.0 mg, 2.5 mg, 3.0 mg, 3.5 mg, or 4.5 mg, twice or three times a day for 12 weeks to Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day
Arm/Group | From PPX ER to PPX ER | From PPX IR to PPX ER
Number analyzed (Participants) | 50 | 53
UPDRS scores on a scale | -2.2 (0.6) | -0.2 (0.6)

19. Secondary Outcome: Percentage of Patients With no Worsening of UPDRS Parts II+III Total Score by More Than 15% From Week 12 to Week 16 (Open-label: Dose Adjustment Phase)
Description: Percentage of patients with no worsening of UPDRS Parts II+III Total Score by more than 15% from week 12 to week 16 (Open-label: Dose Adjustment Phase)
Time Frame: Week 12 to Week 16
Population: Full Analysis Set (FAS 2) for the open-label period
Measure: Number; unit: percentage of participants
Arm/Group | From PPX ER to PPX ER | From PPX IR to PPX ER
Number analyzed (Participants) | 51 | 53
percentage of participants | 78.4 | 83.0

20. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Week 16 Compared to Patient's CGI-I Status at Week 12 (Open-label: Dose Adjustment Phase)
Description: Clinical Global Impression of Improvement (CGI-I) at week 16 compared to patient's CGI-I status at week 12. CGI-I scores ranging from '1' (very much improved) to '7' (very much worse)
Time Frame: Week 12 to Week 16
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Number; unit: percentage of participants
Groups:
- From PPX IR to PPX ER: From Pramipexole IR (tablets of 0.125 mg and 0.5 mg) dose: 0.25 mg, 1.0 mg, 1.5 mg, 2.0 mg, 2.5 mg, 3.0 mg, 3.5 mg, or 4.5 mg, twice or three times a day to Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day
Arm/Group | From PPX ER to PPX ER | From PPX IR to PPX ER
Number analyzed (Participants) | 50 | 53
percentage of participants
  Very much improved | 0.0 | 1.9
  Much improved | 8.0 | 5.7
  Minimally improved | 48.0 | 35.8
  No change | 34.0 | 50.9
  Minimally worse | 10.0 | 5.7

21. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at Week 16 Compared to Patient's PGI-I Status at Week 12 (Open-label: Dose Adjustment Phase)
Description: Patient Global Impression of Improvement (PGI-I) at week 16 compared to patient's PGI-I status at week 12. PGI-I scores ranging from '1' (very much better) to '7' (very much worse).
Time Frame: Week 12 to Week 16
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Number; unit: percentage of participants
Arm/Group | From PPX ER to PPX ER | From PPX IR to PPX ER
Number analyzed (Participants) | 50 | 53
percentage of participants
  Very much better | 2.0 | 3.8
  Much better | 14.0 | 11.3
  A little better | 36.0 | 35.8
  No change | 36.0 | 39.6
  A little worse | 12.0 | 9.4

22. Secondary Outcome: Change From Baseline in UPDRS (Unified Parkinson's Disease Rating Scale) Parts II+III Total Score (Open-label: Maintenance Phase)
Description: as for outcome 1
Time Frame: Baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: UPDRS scores on a scale
Groups:
- Pramipexole ER: Open-Label Phase: Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day during open label period
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
UPDRS scores on a scale | -15.2 (11.1)

23. Secondary Outcome: UPDRS Parts II+III Total Score Responder Rate (at Least 20% Improvement) (Open-label: Maintenance Phase)
Description: as for outcome 13
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Number; unit: percentage of participants
Groups:
- Pramipexole ER: Open-Label Phase: Pramipexole ER (tablets of 0.375 mg and 1.5 mg) dose: 0.375 mg, 0.75 mg, 1.5 mg, 2.25 mg, 3.0 mg, 3.75 mg, or 4.5 mg, once a day during open-label period
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
percentage of participants | 92.0

24. Secondary Outcome: Change From Baseline in Percentage Off-time (Open-label: Maintenance Phase)
Description: as for outcome 2
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: Percentage of off-time
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
Percentage of off-time | -11.6 (22.1)

25. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia (Open-label: Maintenance Phase)
Description: as for outcome 3
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: Percentage of on-time
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
Percentage of on-time | 11.9 (21.1)

26. Secondary Outcome: Change From Baseline in Percentage On-time With Non-troublesome Dyskinesia (Open-label Maintenance Phase)
Description: as for outcome 4
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: Percentage of on-time
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
Percentage of on-time | -0.1 (5.7)

27. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia or With Non-troublesome Dyskinesia (Open-label Maintenance Phase)
Description: as for outcome 5
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: Percentage of on-time
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
Percentage of on-time | 11.8 (21.6)

28. Secondary Outcome: Change From Baseline in Percentage On-time With Troublesome Dyskinesia (Open-label Maintenance Phase)
Description: as for outcome 6
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: Percentage of on-time
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
Percentage of on-time | -0.2 (2.8)

29. Secondary Outcome: Change From Baseline in L-dopa Daily Dose (Open-label Maintenance Phase)
Description: The L-dopa daily dose was recorded in the electronic case report form (eCRF) at each trial visit.
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
mg per day | 10.3 (62.0)

30. Secondary Outcome: Change From Baseline in UPDRS Part I Score (Open-label: Maintenance Phase)
Description: UPDRS Part I ranging from 0 (normal) to 16 (severe). UPDRS Part I measures Mentation, Behavior and Mood
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: UPDRS scores on a scale
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
UPDRS scores on a scale | -0.3 (1.5)

31. Secondary Outcome: Change From Baseline in UPDRS Part II Score (Open-label: Maintenance Phase)
Description: as for outcome 10
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: UPDRS scores on a scale
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
UPDRS scores on a scale | -3.4 (4.2)

32. Secondary Outcome: Change From Baseline in UPDRS Part III Score (Open-label: Maintenance Phase)
Description: UPDRS Part III ranging from 0 (normal) to 108 (severe). UPDRS Part III measures motor symptoms
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Least Squares Mean (Standard Error); unit: UPDRS scores on a scale
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
UPDRS scores on a scale | -11.9 (8.2)

33. Secondary Outcome: Change From Baseline in UPDRS Part IV Score (Open-label: Maintenance Phase)
Description: UPDRS Part IV ranging from 0 (normal) to 23 (severe). UPDRS Part IV measures complications of therapy
Time Frame: baseline and after 64 weeks treatment
Population: Full Analysis Set (FAS 2) for open label period with observed case (OC)
Measure: Mean (Standard Deviation); unit: UPDRS scores on a scale
Arm/Group | Pramipexole ER: Open-Label Phase
Number analyzed (Participants) | 87
UPDRS scores on a scale | -0.6 (1.6)

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication onwards through the observational phase (64 weeks).
Arm/Group | Pramipexole Extended Release Group (PPX ER) | Pramipexole Immediate Release Group (PPX IR)
Serious Adverse Events (participants affected / at risk) | 12/56 | 10/56
Other Adverse Events (participants affected / at risk) | 52/56 | 49/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Extended Release Group (PPX ER) (N=56) | Pramipexole Immediate Release Group (PPX IR) (N=56)
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Delusion (Psychiatric disorders) | 1 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 1
Parkinson's disease (Nervous system disorders) | 1 | 2
Chronic inflammatory polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole Extended Release Group (PPX ER) (N=56) | Pramipexole Immediate Release Group (PPX IR) (N=56)
Nasopharyngitis (Infections and infestations) | 18 | 18
Decreased appetite (Metabolism and nutrition disorders) | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hallucination, visual (Psychiatric disorders) | 7 | 7
Insomnia (Psychiatric disorders) | 4 | 4
Delirium (Psychiatric disorders) | 3 | 0
Somnolence (Nervous system disorders) | 21 | 20
Dyskinesia (Nervous system disorders) | 9 | 4
Dizziness (Nervous system disorders) | 8 | 4
Dizziness postural (Nervous system disorders) | 5 | 3
Sudden onset of sleep (Nervous system disorders) | 3 | 2
Asthenopia (Eye disorders) | 1 | 3
Orthostatic hypotension (Vascular disorders) | 7 | 5
Hypotension (Vascular disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 7 | 12
Nausea (Gastrointestinal disorders) | 8 | 10
Stomatitis (Gastrointestinal disorders) | 6 | 1
Dental caries (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Gastritis (Gastrointestinal disorders) | 1 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Oedema peripheral (General disorders) | 7 | 3
Fall (Injury, poisoning and procedural complications) | 7 | 10
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.